CLINICAL TRIAL: NCT04989114
Title: Effectiveness of Nasal Bubble Continuous Positive Airway Pressure in Reducing Respiratory Distress in Comparison to Standard Care in Children With Bronchiolitis: A Randomized Clinical Trial
Brief Title: Nasal Bubble Continuous Positive Airway Pressure in Reducing Respiratory Distress in Children With Bronchiolitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ameer asadullah gull (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Sponsor-Investigator, ameer asadullah gull, Postgraduate Resident Pediatric Medicine, King Edward Medical University
Organization: King Edward Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 704/RC/KEMU
Record Dates: First submitted 2021-07-14; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Bronchiolitis Acute Viral; Bronchiolitis; Bronchiolitis Acute; Bronchiolitis, Viral; Nasal Continuous Positive Airway Pressure
MeSH Terms: conditions — Bronchiolitis; Bronchiolitis, Viral | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (No Intervention): In this arm, oxygen inhalation will be provided without positive end expiratory pressure
- nasal continuous positive airway pressure (Experimental): In this arm, positive end expiratory pressure will be provided by nasal continuous positive airway pressure
  Interventions: Device: nasal continuous positive airway pressure

INTERVENTIONS:
Device: nasal continuous positive airway pressure — positive end expiratory pressure will be applied by nasal continuous positive airway pressure
  Arms: nasal continuous positive airway pressure

SUMMARY:
This study is designed to assess the effectiveness of nasal continuous positive airway pressure in reducing respiratory distress in children with bronchiolitis

DETAILED DESCRIPTION:
In this study, after taking consent from caretakers, patients of brochiolitis will be randomly assigned to either a standard care group or a nasal continuous positive airway pressure group. Both groups will be followed for respiratory distress. Respiratory distress will be compared by using Seattle sore of respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Children presenting with history of cough, and tachypnea and wheezing on clinical examination

Exclusion Criteria:

* Patients needing mechanical ventilation at the time of admission
* Patients whose caretakers refuse written informed consent
* Patients having consolidation on chest X-Ray

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2020-09-06 (Actual); Primary Completion 2021-09-05 (Estimated); Study Completion 2021-09-05 (Estimated)

PRIMARY OUTCOMES:
reduction in seattle score | after 12 hours
  seattle score will be noted and compared for both groups

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Haroon Hamid, MBBSFCPSFRCS, Principal Investigator — King Edward Medical University
Locations (1):
- Mayo Hospital, Lahore, Punjab Province, Pakistan